CLINICAL TRIAL: NCT07218146
Title: A Randomized, Open-Label, Phase 3 Study of ZL-1310, a DLL3 Antibody-Drug Conjugate (ADC), Compared to Investigator's Choice Therapy in Participants With Relapsed Small Cell Lung Cancer
Brief Title: A Study of ZL-1310 Versus Investigator's Choice of Therapy in Participants With Relapsed Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zai Lab (Shanghai) Co., Ltd. (Industry)
Collaborators: Zai Lab (US) LLC (Industry)
Responsible Party: Sponsor
Organization: Zai Lab (Hong Kong), Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZL-1310-003
Record Dates: First submitted 2025-10-08; First posted 2025-10-20 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): ZL-1310 as a single agent
  Interventions: Drug: ZL-1310
- Arm 2 (Active Comparator): Investigator's Choice of Therapy
  Interventions: Drug: Investigator's Choice of Therapy

INTERVENTIONS:
Drug: ZL-1310 — ZL-1310 as a single-agent
  Arms: Arm 1
Drug: Investigator's Choice of Therapy — Topotecan, Lurbinectedin, or Amrubicin
  Arms: Arm 2

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ZL-1310 compared to Investigator's Choice Therapy in participants with relapsed Small Cell Lung Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years, or considered an adult by local regulations, at the time of consent
* Signed informed consent
* Histologically or cytologically confirmed SCLC. Received 1L platinum-based systemic therapy and had documented disease progression during or after the most recent systemic therapy. Or received 2L tarlatamab is allowed.
* Measurable disease according to RECIST v1.1 as assessed by the investigator.
* Participants with a history of treated and stable or untreated and asymptomatic CNS metastases based on criteria per protocol.
* Adequate organ and marrow function
* Eastern Cooperative Group (ECOG) performance status of 0 or 1
* Life expectancy of at least 3 months
* Participants must be willing to undergo a tumor biopsy or provide archived tumor tissue sample at Screening
* Participants must be willing and able to comply with protocol for the duration of the study

Exclusion Criteria:

* Received more than one line of systemic therapy for Extensive-Stage SCLC.
* Received any prior ADC with topoisomerase 1 inhibitor payload
* Participants with another known malignancy with exceptions defined in the protocol.
* History or suspected ILD/pneumonitis based on criteria per protocol
* Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses.
* Receipt of anti-cancer treatment known to treat cancers within 3 weeks before the first dose of study treatment.
* Prior radiotherapy before study treatment based on criteria per protocol
* Unresolved toxicity of Grade >/= 2 from previous anti-cancer treatment, except for alopecia and skin pigmentation.
* Known infection or active infection defined in the protocol.
* Clinically significant active cardiovascular disease or history of arterial thromboembolic event within 6 months prior to the first dose of study treatment based on criteria per protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2025-11-30 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Confirmed objective response rate (ORR) assessed by Blinded Independent Central Review of ZL-1310 compared to Investigator's Choice Therapy (ICT) | up to 27 months
Overall survival of ZL-1310 compared to Investigator's Choice Therapy (ICT) | up to 27 months

SECONDARY OUTCOMES:
Duration of response (DoR) assessed by BICR and by the investigator per RECIST v1.1 of ZL-1310 compared to Investigator's Choice Therapy (ICT) | up to 27 months
Progression-free survival (PFS) assessed by BICR and by the investigator per RECIST v1.1 of ZL-1310 compared to Investigator's Choice Therapy (ICT) | up to 27 months
Confirmed ORR assessed by the investigator per RECIST v1.1 of ZL-1310 compared to Investigator's Choice Therapy (ICT) | up to 27 months
Time to response (TTR) assessed by BICR and by the investigator per RECIST v1.1 of ZL-1310 compared to Investigator's Choice Therapy (ICT) | up to 27 months
Confirmed CNS response assessed by BICR per Response Assessment in Neuro-Oncology for Brain Metastases (RANO-BM) of ZL-1310 compared to Investigator's Choice Therapy (ICT) | up to 27 months
Occurrence of treatment-emergent adverse events (TEAEs) of ZL-1310 compared to Investigator's Choice Therapy (ICT) | up to 27 months
Changes from baseline in quality of life related parameters of ZL-1310 compared to Investigator's Choice Therapy (ICT) using EQ-5D-5L | up to 27 months
Changes from baseline in quality of life related parameters of ZL-1310 compared to Investigator's Choice Therapy (ICT) using EORTC-QLQ-C30 | up to 27 months
Changes from baseline in quality of life related parameters of ZL-1310 compared to Investigator's Choice Therapy (ICT) using EORTC-QLQ-LC13 | up to 27 months

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Zai Lab Site 02045, Clermont, Florida
  - Zai Lab Site 02031, Orange City, Florida
  - Zai Lab Site 02049, Peoria, Illinois
  - Zai Lab Site 02041, Louisville, Kentucky
  - Zai Lab Site 02003, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No